CLINICAL TRIAL: NCT00498953
Title: Phase I/II Study on Induction Chemotherapy Followed by Chemoradiation With or Without Lapatinib, a Dual EGFR/ErbB2 Kinase Inhibitor, in Patients With Locally Advanced Larynx and Hypopharynx Squamous Cell Carcinoma
Brief Title: Combination Chemotherapy and Radiation Therapy With or Without Lapatinib in Treating Patients With Locally Advanced Cancer of the Larynx or Hypopharynx
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-24051; 2006-002667-33 (EudraCT Number); GSK-EORTC-24051
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Head and Neck Cancer
Keywords: stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin; Cisplatin; Docetaxel; Fluorouracil; Lapatinib; Cytogenetic Analysis; In Situ Hybridization, Fluorescence; In Situ Hybridization; Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction; Immunohistochemistry; Neoadjuvant Therapy; Fluorodeoxyglucose F18; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: docetaxel
Drug: fluorouracil
Drug: lapatinib ditosylate
Genetic: cytogenetic analysis
Genetic: fluorescence in situ hybridization
Genetic: in situ hybridization
Genetic: polymerase chain reaction
Genetic: reverse transcriptase-polymerase chain reaction
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: fludeoxyglucose F 18
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, cisplatin, fluorouracil, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving combination chemotherapy together with radiation therapy, with or without lapatinib, before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed or eliminate the need for surgery.

PURPOSE: This phase I/II trial is studying the side effects and best dose of combination chemotherapy given together with radiation therapy with or without lapatinib and to see how well it works in treating patients with locally advanced cancer of the larynx or hypopharynx.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and recommended dose for phase II of lapatinib ditosylate in patients with locally advanced squamous cell carcinoma of the larynyx or hypopharynx who are concomitantly treated with neoadjuvant induction chemotherapy comprising docetaxel, cisplatin, and fluorouracil, followed by chemoradiotherapy comprising carboplatin and radiotherapy. (Phase I)
* To document the feasibility, in the framework of an organ preservation program, of this regimen in these patients. (Phase II)

Secondary

* To look at the role of PET in patients with N1-3 disease, in terms of PET being used as a reliable method to spare patients from planned neck dissection. (Phase II)

OUTLINE: This is a multicenter, dose-escalation phase I study followed by a randomized phase II study. Patients are stratified by institution and EGFR status (negative vs positive).

* Phase I:

  * Neoadjuvant chemotherapy: Patients receive neoadjuvant chemotherapy comprising docetaxel IV and cisplatin IV on day 1 and fluorouracil IV continuously on days 1-5. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients with a complete or partial response after 4 courses of neoadjuvant chemotherapy proceed to chemoradiotherapy. Patients with less than a partial response after course 2 or course 4 proceed to surgery, including total laryngectomy.
  * Chemoradiotherapy: Within 3 weeks after completion of neoadjuvant chemotherapy, patients undergo radiotherapy on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, and 43-47 and receive carboplatin IV on days 1, 8, 15, 22, 29, 36, and 43.
  * Concurrent lapatinib ditosylate: Patients receive oral lapatinib ditosylate once daily during neoadjuvant chemotherapy, during the break between neoadjuvant chemotherapy and chemoradiotherapy, and during chemoradiotherapy.
* Phase II: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive neoadjuvant chemotherapy and undergo chemoradiotherapy as in phase I.
  * Arm II: Patients receive neoadjuvant chemotherapy and undergo chemoradiotherapy as in phase I. Patients also receive concurrent lapatinib ditosylate as in phase I at the recommended dose determined in phase I.

In both phases, treatment continues in the absence of disease progression or unacceptable toxicity.

Patients with node-positive disease (initially) undergo tumor and blood sample collection for biological studies. Samples are analyzed for ErbB-related activation via immunohistochemistry, in situ hybridization, and PCR/sequencing of genes/proteins, to detect DNA amplification and polysomy (for AKT, ErbB2, EGFR) and genomic losses (for PTEN) via FISH, and the ratio between EGFR and EGFRvIII via QRT-PCR. Patients with node-positive disease undergo at least elective neck dissection to evaluate the negative predictive value of PET scanning.

Patients are followed every 3 months for one year and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed squamous cell carcinoma of the larynx or hypopharynx

  * T3 or T4 disease of the larynx or T2, T3 or T4 disease of the hypopharynx
  * Nodal status must be N0, N1, N2a, N2b, N2c or N3
* Resectable or unresectable disease (Phase I patients only)
* Patient must have tumors amenable to surgery (Phase II patients only)
* No distant metastasis

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin < 1.5 times the upper limit of the normal range
* Alkaline phosphatase and transaminases < 2.5 times the upper limit of the normal range
* Serum creatinine < 1.7 mg/dL
* All patients (male and female) must use effective contraception methods if of reproductive potential (e.g., implants, injectables, combined oral contraceptives, IUDs, sexual abstinence, or vasectomized partner)
* Females must not be pregnant or lactating
* Patients must have normal cardiac function (LVEF assessed by MUGA or ECHO) and clinically satisfactory 12-lead ECG
* No serious cardiac illness or medical condition within the past 6 months including, but not limited to, any of the following:

  * History of documented congestive heart failure
  * High-risk uncontrolled arrhythmias
  * Angina pectoris requiring antianginal medication
  * Clinically significant valvular heart disease
  * Evidence of transmural infarction on ECG
  * Poorly controlled hypertension (e.g., systolic BP > 180 mm Hg or diastolic BP > 100 mm Hg)
* Patients should be able to swallow oral agents
* No current malignancies at other sites with the exception of cone biopsied carcinoma of the cervix and adequately treated basal or squamous cell skin carcinoma or other cancer from which the patient has been disease-free for at least five years
* Absence of any unstable systemic diseases or active uncontrolled infections
* Absence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

PRIOR CONCURRENT THERAPY:

* No other prior therapy for head and neck cancer
* More than 10 days since prior and no concurrent CYP3A4 inducers, including the following:

  * Antibiotics (e.g., all rifamycin class agents [rifampicin, rifabutin, or rifapentine])
  * Anticonvulsants (e.g., phenytoin, carbamezepine, or barbiturates [phenobarbital])
  * Oral glucocorticoids (e.g., cortisone [> 50 mg], hydrocortisone [> 40 mg], prednisone [> 10 mg], methylprednisolone [> 8 mg], or dexamethasone [> 1.5 mg])
  * Antiretrovirals (e.g., efavirenz or nevirapine)
  * Other (hypericum perforatum [St. John's Wort] or modafinil)
* More than 10 days since prior and no concurrent CYP3A4 inhibitors, including the following:

  * Antibiotics (e.g., clarithromycin, erythromycin, or troleandomycin)
  * Antifungals (e.g., itraconazole, ketoconazole, fluconazole [> 150 mg daily], or voriconazole)
  * Antiretrovirals and protease inhibitors (e.g., delavirdine, nelfinavir, amprenavir, ritonavir, indinavir, saquinavir, or lopinavir)
  * Calcium channel blockers (e.g., verapamil or diltiazem)
  * Antidepressants (e.g., nefazodone or fluvoxamine)
  * Gastrointestinal agents (e.g., cimetidine or aprepitant)
  * Other (e.g., grapefruit, grapefruit juice, or camiodarone)
  * Miscellaneous (e.g., antacids [Mylanta, Maalox, Tums, or Rennies], all herbal [bergamottin or glabridin] or dietary supplements)
* Patients may not receive any other anticancer therapy or investigational agents while on study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-05; Primary Completion 2008-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of lapatinib ditosylate (Phase I)
Dose-limiting toxicities of lapatinib ditosylate (Phase I)
Recommended dose of lapatinib ditosylate (Phase I)
Feasibility (Phase II)

SECONDARY OUTCOMES:
Toxicity (Phase II)
Survival with functional larynx (i.e., alive without local progression/relapse, tracheotomy, feeding tube, gastrostomy, or laryngectomy) (Phase II)
Response rate (CR and PR) of neoadjuvant treatment (Phase II)
Overall response rate (Phase II)
Rate of local relapse (Phase II)
Distant metastasis (Phase II)
Overall survival (Phase II)
Predictive value of PET to spare neck dissection in N1-3 patients (Phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Awada, MD, PhD, Study Chair — Jules Bordet Institute
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

REFERENCES:
- [Result] Lalami Y, Specenier PM, Awada A, Lacombe D, Liberatoscioli C, Fortpied C, El-Hariry I, Bogaerts J, Andry G, Langendijk JA, Vermorken JB. EORTC 24051: unexpected side effects in a phase I study of TPF induction chemotherapy followed by chemoradiation with lapatinib, a dual EGFR/ErbB2 inhibitor, in patients with locally advanced resectable larynx and hypopharynx squamous cell carcinoma. Radiother Oncol. 2012 Nov;105(2):238-40. doi: 10.1016/j.radonc.2012.08.006. Epub 2012 Sep 16. PMID 22989664